CLINICAL TRIAL: NCT05950256
Title: Physiological Impact of Surgical Mask and N95 Mask on Obese Operating Room Staff：A Randomized-Controlled Cross-Over Trial
Brief Title: Physiological Impact of Surgical Mask and N95 Mask on Obese Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: KYLL-202306-032
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N95 Respirators

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N95 mask group (Experimental): Continuously wearing N95 mask for 4 hours
  Interventions: Device: N95 mask and surgical mask
- Surgical mask group (Active Comparator): Continuously wearing surgical mask for 4 hours
  Interventions: Device: N95 mask and surgical mask

INTERVENTIONS:
Device: N95 mask and surgical mask — Twenty participants were randomly assigned to the N95 mask group (n=10 ) and the Surgical mask group (n=10 ). The N95 mask group and the Surgical mask group were used in two stages alternately. When the first round of the test was completed and after a 24-hour washing out period, the participants of the Surgical mask group and the N95 respirator group were exchanged for the second round of the test.

SUMMARY:
During the SARS CoV-2 pandemic, in order to reduce the risk of infection among healthcare workers, healthcare workers are usually required to wear N95 masks for extended periods of time in high-risk environments. The long-term use of masks by medical staff has been proven to be related to various symptoms, including headaches, dizziness, facial skin disease symptoms, and other occupational disturbances . Our previous research found that among healthy anesthesiologists with normal weight, wearing a Surgical mask for more than 2h can significantly reduce peripheral blood oxygen saturation (SpO2) and increase respiratory rate (RR). Rebmann et al. investigated the physiological effects of N95 masks on healthcare workers, and the results showed a statistically significant increase in end-tidal CO2 pressure （PetCO2）among 10 intensive care unit nurses who used N95 masks on a 12 hour shift. Recently, it has been confirmed that prolonged use of N95 masks can cause changes in gas exchange, including a decrease in plasma pH and venous partial pressure of oxygen (PvO2), and a slight increase in PetCO2.

Obesity is defined as abnormal or excessive fat accumulation that poses a risk to health and can cause baseline lung function impairment and decreased immune function. According to the standards of the World Health Organization (WHO), people with a body mass index (BMI) greater than 30 kg/m2 are classified as obese. Research shows that obese patients are the population with the highest risk of SARS CoV-2 infection related incidence rate and mortality. Research has shown that healthcare workers who work long hours are more likely to become obese due to changes in body regulation, metabolism, and stress. Long term use of N95 masks by medical staff may lead to a certain degree of insufficient ventilation and/or CO2 re breathing. Obesity itself has a significant impact on the heart and lungs, but the potential physiological effects of long-term wearing of N95 masks on obese healthcare workers have not been studied. The purpose of our study is to determine the abnormal gas exchange and physiological changes of obese doctors and nurses in the operating room who wear Surgical mask and N95 mask for 4 hours.

DETAILED DESCRIPTION:
We plan to recruit 20 non-smoking and healthy obese medical staff, regardless of gender, from the anesthesia doctors and nurses in the operating room, who sign written informed consent forms.

This is a prospective, randomized, cross controlled trial. Develop a sequence number for 20 participants in the order of enrollment. The participants were randomly assigned to the N95 mask group (n=10 cases) and the Surgical mask group (n=10 cases) using the random number method. Before the participants are grouped, group concealment is performed and the random grouping scheme is saved using a shaded envelope. Open the envelopes in the order of the participants joining the group, and determine the grouping situation based on the allocation plan inside the envelopes. The N95 respirator group and the Surgical mask group were used in the two stages of cross operation. When the first round of test was completed and after a 24-hour washing out period, the subjects in the Surgical mask group and the N95 respirator group were exchanged for the second round of test. The steps and methods were the same as those in the first stage.

During the study, each candidate must correctly wear a disposable bandage type medical Surgical mask or a disposable N95 mask. After wearing, it is necessary to check whether it is worn properly and whether there is air leakage. At the beginning of the test, participants are required to avoid using masks for at least 10 minutes, measure their right index finger in a sitting position, and collect baseline (T1) data under normal breathing, including SpO2, Pulse rate (PR), RR, PetCO2, blood pressure (BP). Collect 1ml of venous blood to measure the baseline venous blood gas value.

All subjective sensations were rated using a 10 point VAS digital scale for subjective sensations such as headache, dizziness, difficulty breathing, and facial discomfort. A score of 0 indicates no discomfort, while a score of 10 indicates the most severe imaginable discomfort. Then participants were asked to wear Surgical mask or N95 mask for 4 hours to start medical work. Subsequently, immediately after using masks (T2) and continuously wearing masks for 1 hour (T3), 2 hours (T4), 3 hours (T5), and 4 hours (T6), the above data was collected using the same method. In order to minimize data variability, data was collected twice at each time point and the average was taken. After continuous wear for 4 hours, 1ml of venous blood was taken for blood gas analysis.

If the subject is unable to persist, they can immediately remove the cover and abandon the experiment; Researchers monitored these subjects until symptoms improved. Second round test: After the first round of test is completed, the second round test is conducted after a 24-hour washing period. In the second round of test, the subjects of N95 mask group and Surgical mask group in the first round of test were exchanged, and the test was conducted according to the steps and data collection methods of the first round of test.

ELIGIBILITY:
Inclusion criteria： anesthesiologists or nurses working in the operating room, aged 20-60 years old, body mass index (BMI)>30kg/m2, clearly healthy, and without any history of chronic diseases.

Exclude criteria： recent acute or chronic respiratory disease, recent history of headache and dizziness, pregnancy or lactation, rhinitis, Nasal polyp or poor breathing, facial skin inflammation and skin laxity.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
PvCO2 | 4 hours
  PvCO2 values in venous blood gas after wearing surgical masks or N95 masks for 4 hours

SECONDARY OUTCOMES:
peripheral oxygen saturation (SpO2) | 4 hours
  6 time points before, immediately, 1 hour (h), 2h, 3h and 4h after the continuous wearing of Surgical mask or N95 mask
pulse rate (PR) | 4 hours
  6 time points before, immediately, 1h, 2h, 3h and 4h after the continuous wearing of Surgical mask or N95 mask
PetCO2 | 4 hours
  6 time points before, immediately, 1h, 2h, 3h and 4h after the continuous wearing of Surgical mask or N95 mask
Visual analog scale (VAS) scores | 4 hours
  All sensations were scored by means of a 10-point VAS from 0 (no discomfort) to 10 (worst discomfort imaginable). To minimize variability, data were collected twice at each point in time. To score the subjective discomfort (including dizziness, headache, dyspnea and nasofacial discomfort).
PvCO2 | 0 hours
  PvCO2 in venous blood gas before wearing a mask
PvO2 | 0 hours，4 hours
  PvO2 in venous blood before and after wearing a mask for 4 hours
pH | 0 hours，4 hours
  pH in venous blood before and after wearing a mask for 4 hours
HCO3- | 0 hours，4 hours
  HCO3- in venous blood before and after wearing a mask for 4 hours
systolic pressure | 6 time points before, immediately, 1h, 2h, 3h and 4h after the continuous wearing of Surgical mask or N95 mask
  systolic pressure
diastolic pressure | 6 time points before, immediately, 1h, 2h, 3h and 4h after the continuous wearing of Surgical mask or N95 mask
  diastolic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shaozhong Yang, Doctor, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
After the research is completed, share research data, research plans, statistical analysis plans, informed consent forms, and other data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2024- December 2024
Access Criteria: Network access or email
URL: http://www.medresman.org.cn/uc/sindex.aspx

REFERENCES:
- [Result] Luo C, Yao L, Zhang L, Yao M, Chen X, Wang Q, Shen H. Possible Transmission of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in a Public Bath Center in Huai'an, Jiangsu Province, China. JAMA Netw Open. 2020 Mar 2;3(3):e204583. doi: 10.1001/jamanetworkopen.2020.4583. Erratum In: JAMA Netw Open. 2020 Aug 3;3(8):e2017413. doi: 10.1001/jamanetworkopen.2020.17413. PMID 32227177
- [Result] O'Hara LM, Thom KA, Preas MA. Update to the Centers for Disease Control and Prevention and the Healthcare Infection Control Practices Advisory Committee Guideline for the Prevention of Surgical Site Infection (2017): A summary, review, and strategies for implementation. Am J Infect Control. 2018 Jun;46(6):602-609. doi: 10.1016/j.ajic.2018.01.018. Epub 2018 Mar 7. PMID 29525367
- [Result] Scheid JL, Lupien SP, Ford GS, West SL. Commentary: Physiological and Psychological Impact of Face Mask Usage during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Sep 12;17(18):6655. doi: 10.3390/ijerph17186655. PMID 32932652
- [Result] Yang S, Fang C, Liu X, Liu Y, Huang S, Wang R, Qi F. Surgical Masks Affect the Peripheral Oxygen Saturation and Respiratory Rate of Anesthesiologists. Front Med (Lausanne). 2022 Apr 14;9:844710. doi: 10.3389/fmed.2022.844710. eCollection 2022. PMID 35492371
- [Result] Rebmann T, Carrico R, Wang J. Physiologic and other effects and compliance with long-term respirator use among medical intensive care unit nurses. Am J Infect Control. 2013 Dec;41(12):1218-23. doi: 10.1016/j.ajic.2013.02.017. Epub 2013 Jun 12. PMID 23768438
- [Result] Shechtman L, Ben-Haim G, Ben-Zvi I, Steel L, Ironi A, Huszti E, Chatterji S, Levy L. Physiological Effects of Wearing N95 Respirator on Medical Staff During Prolong Work Hours in Covid-19 Departments. J Occup Environ Med. 2022 Jun 1;64(6):e378-e380. doi: 10.1097/JOM.0000000000002542. Epub 2022 May 4. PMID 35543650
- [Result] Zhou Y, Chi J, Lv W, Wang Y. Obesity and diabetes as high-risk factors for severe coronavirus disease 2019 (Covid-19). Diabetes Metab Res Rev. 2021 Feb;37(2):e3377. doi: 10.1002/dmrr.3377. Epub 2020 Jul 20. PMID 32588943
- [Result] Luckhaupt SE, Cohen MA, Li J, Calvert GM. Prevalence of obesity among U.S. workers and associations with occupational factors. Am J Prev Med. 2014 Mar;46(3):237-48. doi: 10.1016/j.amepre.2013.11.002. PMID 24512862
- [Result] Sharma SV, Upadhyaya M, Karhade M, Baun WB, Perkison WB, Pompeii LA, Brown HS, Hoelscher DM. Are Hospital Workers Healthy?: A Study of Cardiometabolic, Behavioral, and Psychosocial Factors Associated With Obesity Among Hospital Workers. J Occup Environ Med. 2016 Dec;58(12):1231-1238. doi: 10.1097/JOM.0000000000000895. PMID 27930484
- [Result] Dixon AE, Peters U. The effect of obesity on lung function. Expert Rev Respir Med. 2018 Sep;12(9):755-767. doi: 10.1080/17476348.2018.1506331. Epub 2018 Aug 14. PMID 30056777
- [Derived] Fang C, Ba Y, Gao Y, Liu Y, Yang S. Physiological impact of surgical masks and N95 masks on obese operating room staff. Sci Rep. 2025 Feb 24;15(1):6533. doi: 10.1038/s41598-025-91578-9. PMID 39994350